CLINICAL TRIAL: NCT02777840
Title: High Flow Oxygen With THRIVE Gives Better Oxygenation in Rapid Sequence Induction Patients
Acronym: THRIVE/RSI 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15/LO/0277
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: High Flow Oxygen in Rapid Sequence Induction; Airway Morbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Face mask group (Active Comparator): Patients will be given oxygen via face mask as per routine practice, blood gas sample taken after airway is secured, heart rate of anaesthetist monitored and time for desaturation noted.
  Interventions: Device: face mask oxygen
- THRIVE group (Active Comparator): Patients will be given oxygen via high flow oxygen in Optiflo, blood gas sample taken after airway is secured, heart rate of anaesthetist monitored and time for desaturation noted.
  Interventions: Device: High flow oxygen

INTERVENTIONS:
Device: face mask oxygen — oxygen given by face mask as per routine practice
  Arms: Face mask group
Device: High flow oxygen — High flow oxygen given via optiflo machine / device
  Arms: THRIVE group

SUMMARY:
High flow oxygen results in better oxygenation in emergency cases needing rapid sequence induction for anaesthesia. Secondary outcome measure is time for any desaturation.

DETAILED DESCRIPTION:
The investigators intend to do the study using high flow oxygen for all emergency cases needing rapid sequence induction. As part of the study the Investigators will measure the oxygen levels in the blood gas sample of the patient and the heart rate of anesthetist in charge of the airway management. After the airway is secured the time for desaturation will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Emergency patients needing rapid sequence induction for surgery
* ≥ 16 years
* Able to give consent

Exclusion Criteria:

* Patients age under 16 years
* Inability to give consent
* Severe respiratory disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Oxygen levels in blood gas sample | intraoperative
  Oxygen levels in blood gas sample after the airway is secured

SECONDARY OUTCOMES:
time to desaturation | intraoperative or 10 minutes after intubation
  after airway is secured time will be noted for oxygen levels to fall to 92% before the ventilation is started.
heart rate of anaesthetist performing the intubation | During the process of induction of anaesthesia and intubation upto 5 minutes post intubation

CONTACTS AND LOCATIONS:
Overall Officials: Fauzia Mir, Principal Investigator — St Georges hospital NHS trust
Locations (1):
- St Georges Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
As per guidelines